CLINICAL TRIAL: NCT02188108
Title: Validation of the Wisconsin Stone-QOL, a Quality of Life Survey for Kidney Stone Formers
Brief Title: Validation of the Wisconsin Stone-QOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: University of Florida (Other); University of California, San Diego (Other); University of North Carolina (Other); Dartmouth College (Other); The Cleveland Clinic (Other); University of British Columbia (Other); University of Texas (Other); University of California, Davis (Other); University of California, Irvine (Other); University of California, San Francisco (Other); University of Washington (Other); Penn State University (Other); McGill University (Other); University of Pittsburgh (Other); Université de Montréal (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2014-0062; UW QOL (Other: Study Team); A539998 (Other: UW Madison); SMPH\VOLUNTEER STAFF\UROLOGY (Other: UW Madison); Protocol Version 1/19/2018 (Other: UW Madison)
Record Dates: First submitted 2014-07-07; First posted 2014-07-11 (Estimated); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Urolithiasis; Nephrolithiasis; Kidney Stones
Keywords: quality of life; QOL; urolithiasis; nephrolithiasis; kidney stones; patient-reported outcomes
MeSH Terms: conditions — Urolithiasis; Nephrolithiasis; Kidney Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Survey (Experimental): Wisconsin Stone-QOL survey. Patients with kidney stones or a history thereof will complete a kidney stone-specific health-related survey at enrollment and post-enrollment at 3 months, 12 months, 24 months, and 36 months.
  Interventions: Other: Wisconsin Stone-QOL survey

INTERVENTIONS:
Other: Wisconsin Stone-QOL survey — Patients will complete a health-related quality of life survey at multiple time points at enrollment and at multiple time points thereafter.

SUMMARY:
The overall purpose of this study is to evaluate criterion-related validity of a newly-developed disease-specific instrument to assess the health-related quality of life (HRQOL) of patients who have had kidney stones. Specific aims of this study are:

1. Aim 1. Evaluate the population/external validity (generalizability) of the Wisconsin Stone-QOL by answering the question, "Is the Wisconsin Stone-QOL useful for assessing the HRQOL of patients who form kidney stones from a broad region of North America?"
2. Aim 2. Assess the ability of the Wisconsin Stone-QOL to detect changes within patients related to stone interventions and other disease-specific outcomes by answering the question, "Is the Wisconsin Stone-QOL sensitive to changes in stone-related outcomes within individuals?"

DETAILED DESCRIPTION:
The Wisconsin Stone-QOL was developed as the only known HRQOL instrument designed specifically for patients with kidney stones. Its development has been published. Internal and other validity tests on the instrument have been conducted and reported. Further validity testing of the instrument is needed to confirm its broader utility in the context of surgical and medical management of patients with kidney stones.

Upon enrollment at each site, patients will be asked to complete a medical history form and the Wisconsin Stone-QOL. To supplement the information provided in the medical history forms, patients' medical records will be reviewed in order to collect and enter approved data into a spreadsheet. Further patient interventions include completion of the Wisconsin Stone-QOL at 3 months, 12 months, 24 months, and 36 months post-enrollment. These post-enrollment surveys will usually be mailed to patients to the addresses they provide. Alternatively, patients may be provided the surveys at a urology encounter if it falls on or near the intervention time points. At each time point, patients' medical records will also be searched to document any changes in the data entered at enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of kidney stones, either in the past or currently
* 18 years of age or older

Exclusion Criteria:

* Under 18 years of age
* No previous or current diagnosis of kidney stones

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3299 (Actual)
Dates: Start 2014-07; Primary Completion 2022-05-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Patients' self-reported health-related quality of life (HRQOL) | Enrollment
  Change in HRQOL from baseline to follow-up time points will be assessed

SECONDARY OUTCOMES:
Patients' self-reported quality of life | 3 months

OTHER OUTCOMES:
Patients' self-reported quality of life | 12 months
Patients' self-reported quality of life | 24 months
Patients' self-reported quality of life | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Kristina L Penniston, PhD, Principal Investigator — University of Wisconsin Department of Urology, School of Medicine & Public Health; Stephen Y Nakada, MD, Principal Investigator — University of Wisconsin Department of Urology, School of Medicine & Public Health
Locations (1):
- University of Wisconsin-Madison Department of Urology, School of Medicine & Public Heatlh, Madison, Wisconsin, United States

REFERENCES:
- [Background] Penniston KL, Nakada SY. Health related quality of life differs between male and female stone formers. J Urol. 2007 Dec;178(6):2435-40; discussion 2440. doi: 10.1016/j.juro.2007.08.009. Epub 2007 Oct 15. PMID 17937947
- [Background] Penniston KL, Nakada SY. Development of an instrument to assess the health related quality of life of kidney stone formers. J Urol. 2013 Mar;189(3):921-30. doi: 10.1016/j.juro.2012.08.247. Epub 2012 Sep 24. PMID 23017521
- [Background] Ahmad TR, Tzou DT, Usawachintachit M, Reliford-Titus S, Wu C, Goodman J, Antonelli JA, Viprakasit DP, Averch TD, Sivalingam S, Chew BH, Bird VG, Pais VM Jr, Streeper NM, Sur RL, Nakada SY, Penniston KL, Chi T. Low Income and Nonwhite Race are Strongly Associated with Worse Quality of Life in Patients with Nephrolithiasis. J Urol. 2019 Jul;202(1):119-124. doi: 10.1097/JU.0000000000000233. Epub 2019 Jun 7. PMID 30865567
- [Background] Raffin EP, Penniston KL, Antonelli JA, Viprakasit DP, Averch TD, Bird VG, Chew BH, Sivalingam S, Sur RL, Nakada SY, Pais VM Jr. The Effect of Thiazide and Potassium Citrate Use on the Health Related Quality of Life of Patients with Urolithiasis. J Urol. 2018 Dec;200(6):1290-1294. doi: 10.1016/j.juro.2018.06.023. Epub 2018 Jun 18. PMID 29913138
- [Background] Stern KL, Gao T, Antonelli JA, Viprakasit DP, Averch TD, Chi T, Chew BH, Bird VG, Pais VM Jr, Streeper NM, Sur RL, Nakada SY, Penniston KL, Sivalingam S. Association of Patient Age and Gender with Kidney Stone Related Quality of Life. J Urol. 2019 Aug;202(2):309-313. doi: 10.1097/JU.0000000000000291. Epub 2019 Jul 8. PMID 31026215
- [Background] Atalay HA, Ulker V, Canat L, Ozer M, Can O, Penniston KL. Validation of the Turkish version of the Wisconsin stone-quality of life questionnaire. Turk J Urol. 2018 Mar 16;45(2):118-123. doi: 10.5152/tud.2018.35305. Print 2019 Mar. PMID 29799402
- [Background] Penniston KL, Antonelli JA, Viprakasit DP, Averch TD, Sivalingam S, Sur RL, Pais VM Jr, Chew BH, Bird VG, Nakada SY. Validation and Reliability of the Wisconsin Stone Quality of Life Questionnaire. J Urol. 2017 May;197(5):1280-1288. doi: 10.1016/j.juro.2016.11.097. Epub 2016 Nov 23. PMID 27889419
- [Background] Streeper NM, Wertheim ML, Nakada SY, Penniston KL. Cystine Stone Formers Have Impaired Health-Related Quality of Life Compared with Noncystine Stone Formers: A Case-Referent Study Piloting the Wisconsin Stone Quality of Life Questionnaire Among Patients with Cystine Stones. J Endourol. 2017 Apr;31(S1):S48-S53. doi: 10.1089/end.2016.0564. Epub 2016 Nov 8. PMID 27717296